CLINICAL TRIAL: NCT01700816
Title: Usefulness of Bright Light Therapy in the Prevention of Delirium in Patients Undergoing Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Prevention of Delirium After Bone Marrow Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low incidence of delirium.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Carlos Fernandez-Robles, Principal Investigator, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2010P002801
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Delirium
Keywords: Delirium; Hematopoietic stem cell transplantation; Bone marrow transplantation; Bright Light Therapy
MeSH Terms: conditions — Delirium | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bright light therapy (Experimental): 2500 Lux gaze directed every morning from 8 am until 8:30 am
  Interventions: Device: Bright light therapy
- Sham light (Placebo Comparator): <1000 Lux gaze directed every morning from 8 am until 8:30 am
  Interventions: Device: Sham light

INTERVENTIONS:
Device: Bright light therapy — The light box will be placed vertically on a patient table or bed side 2.5 feet away from the user's eyes daily from 8 am to 8:30 am.
  Other Names: DL930 Day-Light Classic by Uplift Technologies Inc.
  Arms: Bright light therapy
Device: Sham light — The light box will be placed vertically on a patient table or bed side 2.5 feet away from the user's eyes daily from 8 am to 8:30 am.
  Other Names: DL930 Day-Light Classic Uplift Tecnologies placebo box
  Arms: Sham light

SUMMARY:
The purpose of this study is to find out if using bright light sessions during bone marrow transplant can prevent people from developing confusion also known as delirium.

DETAILED DESCRIPTION:
This is a pilot, double blind randomized study conducted in patients scheduled to undergo bone marrow transplant at the Massachusetts General Hospital. The goal of this study is to look at the usefulness of bright light therapy in the prevention of delirium in a population at high risk for developing this condition.

Delirium can develop in up to half of the people that undergo bone marrow transplant. Symptoms include changes in level of alertness, confusion, and temporary problems with memory and attention. In severe cases, it can be accompanied by agitation, paranoia(overly suspicious), and hallucinations(seeing or hearing things that are not really there).

Bright light uses no medication and is often used to treat seasonal affective depression and multiple sleep disorders. The light boxes are portable and are placed in front of individuals for about 30 minutes every day.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Male or female
* Patients scheduled to undergo HSCT
* English speaking

Exclusion Criteria:

* Previous history of bipolar affective disorder
* On-going delirium
* History of substance abuse/dependence within 6 months prior to HSCT
* History of invasive melanoma. Patients with a history of basal cell carcinoma, melanoma in situ, or squamous cell carcinoma are permitted to enroll if the lesion(s) have been excised with negative margins
* History of medical/dermatological conditions that make skin especially sensitive to light,such as systemic lupus erythematosus (SLE) and/or porphyria
* Eye condition that makes eyes vulnerable to light damage
* Concomitant use of medications that increase sensitivity to sunlight, such as the herbal supplement St. John's Wort
* Established primary insomnia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernandez-Robles, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirshner HS. Delirium: a focused review. Curr Neurol Neurosci Rep. 2007 Nov;7(6):479-82. doi: 10.1007/s11910-007-0074-7. PMID 17999893
- [Background] Minden SL, Carbone LA, Barsky A, Borus JF, Fife A, Fricchione GL, Orav EJ. Predictors and outcomes of delirium. Gen Hosp Psychiatry. 2005 May-Jun;27(3):209-14. doi: 10.1016/j.genhosppsych.2004.12.004. PMID 15882768
- [Background] Inouye SK, Schlesinger MJ, Lydon TJ. Delirium: a symptom of how hospital care is failing older persons and a window to improve quality of hospital care. Am J Med. 1999 May;106(5):565-73. doi: 10.1016/s0002-9343(99)00070-4. PMID 10335730
- [Background] Fricchione GL, Nejad SH, Esses JA, Cummings TJ Jr, Querques J, Cassem NH, Murray GB. Postoperative delirium. Am J Psychiatry. 2008 Jul;165(7):803-12. doi: 10.1176/appi.ajp.2008.08020181. No abstract available. PMID 18593786
- [Background] Hshieh TT, Fong TG, Marcantonio ER, Inouye SK. Cholinergic deficiency hypothesis in delirium: a synthesis of current evidence. J Gerontol A Biol Sci Med Sci. 2008 Jul;63(7):764-72. doi: 10.1093/gerona/63.7.764. PMID 18693233
- [Background] Kalisvaart KJ, de Jonghe JF, Bogaards MJ, Vreeswijk R, Egberts TC, Burger BJ, Eikelenboom P, van Gool WA. Haloperidol prophylaxis for elderly hip-surgery patients at risk for delirium: a randomized placebo-controlled study. J Am Geriatr Soc. 2005 Oct;53(10):1658-66. doi: 10.1111/j.1532-5415.2005.53503.x. PMID 16181163
- [Background] Prakanrattana U, Prapaitrakool S. Efficacy of risperidone for prevention of postoperative delirium in cardiac surgery. Anaesth Intensive Care. 2007 Oct;35(5):714-9. doi: 10.1177/0310057X0703500509. PMID 17933157
- [Background] Liptzin B, Laki A, Garb JL, Fingeroth R, Krushell R. Donepezil in the prevention and treatment of post-surgical delirium. Am J Geriatr Psychiatry. 2005 Dec;13(12):1100-6. doi: 10.1176/appi.ajgp.13.12.1100. PMID 16319303
- [Background] Sampson EL, Raven PR, Ndhlovu PN, Vallance A, Garlick N, Watts J, Blanchard MR, Bruce A, Blizard R, Ritchie CW. A randomized, double-blind, placebo-controlled trial of donepezil hydrochloride (Aricept) for reducing the incidence of postoperative delirium after elective total hip replacement. Int J Geriatr Psychiatry. 2007 Apr;22(4):343-9. doi: 10.1002/gps.1679. PMID 17006875
- [Background] Leung JM, Sands LP, Rico M, Petersen KL, Rowbotham MC, Dahl JB, Ames C, Chou D, Weinstein P. Pilot clinical trial of gabapentin to decrease postoperative delirium in older patients. Neurology. 2006 Oct 10;67(7):1251-3. doi: 10.1212/01.wnl.0000233831.87781.a9. Epub 2006 Aug 16. PMID 16914695
- [Background] Tabet N, Howard R. Non-pharmacological interventions in the prevention of delirium. Age Ageing. 2009 Jul;38(4):374-9. doi: 10.1093/ageing/afp039. Epub 2009 May 21. PMID 19460856
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Lipowski ZJ. Delirium (acute confusional states). JAMA. 1987 Oct 2;258(13):1789-92. PMID 3625989
- [Background] Shigeta H, Yasui A, Nimura Y, Machida N, Kageyama M, Miura M, Menjo M, Ikeda K. Postoperative delirium and melatonin levels in elderly patients. Am J Surg. 2001 Nov;182(5):449-54. doi: 10.1016/s0002-9610(01)00761-9. PMID 11754849
- [Background] McIntyre IM, Norman TR, Burrows GD, Armstrong SM. Human melatonin suppression by light is intensity dependent. J Pineal Res. 1989;6(2):149-56. doi: 10.1111/j.1600-079x.1989.tb00412.x. PMID 2915324
- [Background] Petterborg LJ, Kjellman BF, Thalen BE, Wetterberg L. Effect of a 15 minute light pulse on nocturnal serum melatonin levels in human volunteers. J Pineal Res. 1991 Jan;10(1):9-13. doi: 10.1111/j.1600-079x.1991.tb00003.x. PMID 2056432
- [Background] Fortuyn HD, Schoemaker J. Treatment of delirium with phototherapy: a case report. Eur Psychiatry. 1997;12(7):367-8. doi: 10.1016/s0924-9338(97)80007-7. PMID 19698553
- [Background] Schmitz M, Frey R, Pichler P, Ropke H, Anderer P, Saletu B, Rudas S. Sleep quality during alcohol withdrawal with bright light therapy. Prog Neuropsychopharmacol Biol Psychiatry. 1997 Aug;21(6):965-77. doi: 10.1016/s0278-5846(97)00092-4. PMID 9380792
- [Background] Taguchi T, Yano M, Kido Y. Influence of bright light therapy on postoperative patients: a pilot study. Intensive Crit Care Nurs. 2007 Oct;23(5):289-97. doi: 10.1016/j.iccn.2007.04.004. Epub 2007 Aug 9. PMID 17692522
- [Background] Beglinger LJ, Duff K, Van Der Heiden S, Parrott K, Langbehn D, Gingrich R. Incidence of delirium and associated mortality in hematopoietic stem cell transplantation patients. Biol Blood Marrow Transplant. 2006 Sep;12(9):928-35. doi: 10.1016/j.bbmt.2006.05.009. PMID 16920558
- [Background] Fann JR, Roth-Roemer S, Burington BE, Katon WJ, Syrjala KL. Delirium in patients undergoing hematopoietic stem cell transplantation. Cancer. 2002 Nov 1;95(9):1971-81. doi: 10.1002/cncr.10889. PMID 12404292
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Reitan RM. Validity of the Trail Making test as an indicator of organic brain damage. Perceptual and Motor Skills 8: 271-276, 1958.
- [Background] Derogatis LR, Savitz, KL. The SCL-90-R and the Brief Symptom Inventory (BSI) in Primary Care In: M.E.Maruish, ed. Handbook of psychological assessment in primary care settings 236: 297,334, 2000. Mahwah, NJ: Lawrence Erlbaum Associates.
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Breitbart W, Rosenfeld B, Roth A, Smith MJ, Cohen K, Passik S. The Memorial Delirium Assessment Scale. J Pain Symptom Manage. 1997 Mar;13(3):128-37. doi: 10.1016/s0885-3924(96)00316-8. PMID 9114631
- [Background] Lewy AJ, Wehr TA, Goodwin FK, Newsome DA, Markey SP. Light suppresses melatonin secretion in humans. Science. 1980 Dec 12;210(4475):1267-9. doi: 10.1126/science.7434030.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bright Light Therapy | Sham Light
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright Light Therapy | Sham Light | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.84) | 53.1 (14.15) | 53.2 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 18 | 10 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Information not provided during interviews by all participants
  Participants
    Non Hispanic White: number analyzed (Participants) | 18 | 17 | 35
    Non Hispanic White | 16 | 17 | 33
    Hispanic or Latino: number analyzed (Participants) | 18 | 17 | 35
    Hispanic or Latino | 1 | 0 | 1
    Asian: number analyzed (Participants) | 18 | 17 | 35
    Asian | 1 | 0 | 1
Marital Status [Count of Participants; unit: Participants] — Population: Information not provided during interviews by all participants
  Participants
    Married/Partnered: number analyzed (Participants) | 17 | 17 | 34
    Married/Partnered | 12 | 13 | 25
    Single/Divorced/Widowed: number analyzed (Participants) | 17 | 17 | 34
    Single/Divorced/Widowed | 5 | 4 | 9
Highest Education Level [Count of Participants; unit: Participants] — Population: Information not provided during interviews by all participants
  Participants
    11th grade or less: number analyzed (Participants) | 17 | 15 | 32
    11th grade or less | 1 | 0 | 1
    High School degree/GED | 2 | 6 | 8
    Some College | 2 | 2 | 4
    Completed College | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Delirium Based on Meeting Criteria on the Delirium Rating Scale and/or Memorial Delirium Assessment Scale
Description: Monday, Wednesday, and Friday assessments will begin after beginning light therapy and include the Delirium Rating Scale-Revised-98 (DRS-98)and Memorial Delirium Assessment Scale (MDAS)
Time Frame: From hospital admission until the date of first documented delirium, assessed up to 28 days post-transplant
Population: Only 20 bright light therapy and 18 sham light participants were analyzed because 2 participants (one from each arm) only had one assessment. Consequently, no change could be documented to analyze change of delirium scales. They did not drop out; they just completed their transplant before more data could be gathered.
Measure: Count of Participants; unit: Participants
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

2. Secondary Outcome: Severity of Delirium Episodes: Memorial Delirium Assessment Scale (MDAS)
Description: Monday, Wednesday, and Friday assessments of the Memorial Delirium Assessment Scale (MDAS); Patients will receive assessments after beginning light therapy until day 28 post-transplant or discharge, whichever comes first.
  10 item scale Items are rated on a four-point scale from 0 (none) to 3 (severe) depending on the level of impairment, rendering a maximum possible score of 30.
  A score of 13 has been recommended as a cut-off for establishing the diagnosis of delirium
Time Frame: From first documented episode of delirium until discharge from the hospital, assessed up to 28 days post-transplant
Population: Only one case of delirium developed, and only an MDAS score was collected for this participant.
Measure: Number; unit: units on a scale
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 1 | 0
units on a scale | 18 |

3. Secondary Outcome: Average Dose of Antipsychotic Medications Required to Manage Delirium
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: Only one case of delirium developed, and we did not collect data on antipsychotic medication use for this one participant.
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: One participant in the sham light arm was missing date of discharge, so only 18 hospital lengths of stay were able to be calculated in that arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 21 | 18
days | 18 [17 to 21] | 18.5 [15 to 22]

5. Secondary Outcome: Sodium (Na), Potassium (K), Chloride (Cl), and Carbon Dioxide (CO2)
Description: Lab values at latest available follow-up date per participant. These tests are performed as part of routine clinical care on patients undergoing HSCT (Hematopoietic Stem Cell Transplantation).
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: 8 participants were missing lab data in the bright light group, and 7 participants were missing lab data in the sham light group
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
mmol/L
  Sodium (Na) | 139 [137 to 139] | 138.0 [136.0 to 140.5]
  Potassium (K) | 3.6 [3.5 to 3.8] | 3.80 [3.45 to 4.30]
  Chloride (Cl) | 105 [103 to 105] | 103.0 [102.0 to 106.5]
  Carbon Dioxide (CO2) | 24.9 [24.6 to 26.6] | 25.10 [23.40 to 26.55]

6. Secondary Outcome: Serum Creatinine and Blood Urea Nitrogen (BUN)
Description: Lab values at latest available follow-up date per participant. These tests are performed as part of routine clinical care on patients undergoing HSCT.
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
mg/dl
  Serum Creatinine | 0.66 [0.54 to 0.84] | 0.75 [0.47 to 0.84]
  Blood Urea Nitrogen (BUN) | 9 [6 to 12] | 8.5 [4.5 to 10.5]

7. Secondary Outcome: Red Blood Cells (RBC)
Description: as for outcome 6
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: M/uL
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
M/uL | 3.21 [2.88 to 3.31] | 2.93 [2.80 to 3.16]

8. Secondary Outcome: White Blood Cells (WBC)
Description: as for outcome 6
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: K/uL
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
K/uL | 2.30 [2.10 to 4.00] | 4.75 [1.55 to 7.40]

9. Secondary Outcome: Hemoglobin (HGB)
Description: as for outcome 6
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
g/dl | 9.70 [8.90 to 10.20] | 9.55 [8.85 to 9.90]

10. Secondary Outcome: Hematocrit (HCT)
Description: as for outcome 6
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: volume percentage (vol%) of red blood ce
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
volume percentage (vol%) of red blood ce | 28.20 [25.20 to 29.90] | 26.70 [25.70 to 28.65]

11. Secondary Outcome: Platelet Count
Description: as for outcome 6
Time Frame: From admission to hospital to discharge, an expected average of 28 days post-transplant
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: thousand cells/uL
Arm/Group | Bright Light Therapy | Sham Light
Number analyzed (Participants) | 13 | 12
thousand cells/uL | 39 [33 to 94] | 33.5 [24.5 to 47.5]

ADVERSE EVENTS:
Time Frame: 28 days post-transplant or discharge, whichever comes first
Arm/Group | Bright Light Therapy | Sham Light
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No